CLINICAL TRIAL: NCT05655078
Title: Hemithoracic Irradiation With Proton Therapy in Malignant Pleural Mesothelioma
Acronym: HIT-Meso
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Asthma + Lung UK (Unknown); Mesothelioma UK (Unknown); University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/148232; MCTA22F\7 (Other Grant/Funding Number: Asthma _ Lung UK)
Record Dates: First submitted 2022-11-11; First posted 2022-12-16 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Proton beam therapy
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Proton Therapy

STUDY DESIGN:
Intervention Model Description: Control arm (standard of care) vs experimental arm (proton beam therapy) in 1:1 randomisation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): MPM participants who are on the standard of care watch and wait approach i.e. immediate treatment not suitable. Participants will have follow-up for 2 years (3 monthly in year 1, 4 monthly in year 2).
- Proton beam therapy (Experimental): MPM participants to receive 5 weeks of proton beam therapy to the hemithorax. Following completion of treatment participants will have follow-up at the referring centre for 2 years (3 monthly in year 1, 4 monthly in year 2).
  Interventions: Radiation: Proton beam therapy

INTERVENTIONS:
Radiation: Proton beam therapy — 5 weeks (Mon-Fri) of proton beam treatment to the hemithorax to a dose of 50Gy in 25 fractions with a boost to 60Gy for the visible tumour (gross tumour volume-GTV).
  Arms: Proton beam therapy

SUMMARY:
Phase III randomised-controlled trial for patients with unilateral malignant pleural mesothelioma (MPM).

DETAILED DESCRIPTION:
Study design: Randomised phase III clinical trial for patients with unilateral MPM.

Primary endpoint: Progression free survival (PFS) and overall survival (OS), defined as the time from randomisation to the date of progression and death from any cause.

Secondary Endpoints: Safety and Tolerability, Health related Quality of Life (QOL): EuroQoL EQ-5D-3L, Locoregional Control.

Randomisation and stratification: 1:1 randomisation. Patients with be stratified for histology (epithelioid versus non-epithelioid), potential PBT centre (UCLH or The Christie)

, laterality (left or right sided) and time since diagnosis (<1 year or > 1 year)

Treatment:

Experimental Arm: Patients in the experimental arm will receive PBT to the hemithorax to a dose of 50Gy in 25 fractions with a boost to 60Gy for the visible tumour (gross tumour volume-GTV). Treatment is given daily Monday-Friday over 5 weeks. Following completion of treatment in the experimental arm patients will have 2 years of follow-up from time of randomisation at the local recruiting/referring centre.

Control Arm:

The patients in the control arm would be under standard of care surveillance i.e. "watch and wait", with no treatment or other intervention. Patients will have 2 years of follow-up from time of randomisation at the local recruiting/referring centre. If the disease progresses, the patient will receive SOC treatment i.e. immunotherapy with nivolumab and ipilimumab, or chemotherapy at the clinician's discretion.

Statistical analysis plan:

The sample size is 148 patients (74 patients per arm). This is to detect a OS hazard ratio of 0.58, equivalent to an improvement in 2-year OS from 30% to 50%, with 85% power and 5% two-sided alpha. Recruitment to complete in 3 years across 20 UK centres with 2 years of additional follow-up and up to 5% dropout. Interim analyses for OS efficacy will be performed when 50, 75 and 110 patients have been randomised at around 1.5, 2.0 and 2.5 years respectively. Using a fixed-sequence approach, a difference for OS will only be tested if the co-primary endpoint of PFS is statistically significant (p<0.05); N=148 will provide >85% power to detect a PFS hazard ratio of 0.58 accounting for up to 10% dropout.

ELIGIBILITY:
Inclusion criteria:

* Patients ≥18 years of age, with biopsy confirmed MPM and histological subtyping (epithelioid or non-epithelioid)
* N0 or N1 and M0 disease
* Written informed consent
* Patient and local/regional MDT opt for active surveillance and deferral of SACT until clinical or radiological progression
* WHO Performance Status 0-1
* Disease confined to one hemithorax based on CT assessment
* Adequate pulmonary function

  * ≥ 40% predicted post-FEV1;
  * ≥ 40% predicted DLCO/TLCO
* Agreement to travel to either proton beam therapy centres (i.e. UCLH or The Christie) if randomised to arm 2
* Agreement to be followed up at a local HIT-Meso trial site
* Patient likely able to complete PBT planning based on local assessment

Exclusion criteria:

* Presence of metastatic or contralateral disease
* Cytological diagnosis and/or undetermined histological subtype
* Prior thoracic radiotherapy, chemotherapy, immunotherapy for MPM
* Prior radical surgery for MPM (extrapleural pneumonectomy or extended pleurectomy decortication or pleurectomy decortication)
* Initial systemic therapy or surgery is required and the patient and local/regional MDT do not opt for active surveillance
* Involvement of contralateral or supraclavicular lymph nodes
* T4 disease with invasion of the myocardium
* N2 and/or M1 disease
* Presence of new effusion that is not amenable to drainage
* WHO Performance Status ≥ 2
* Women who are pregnant or breast feeding
* Current or previous malignant disease which may impact on the patient's life expectancy
* Patient fitted with a pacemaker or implantable cardioverter-defibrillator (ICD)\
* Diagnosis of clinically significant interstitial lung disease (ILD), excluding mild fibrosis or incidental findings
* Chronic non-malignant disease with an estimated three-year survival rate of less than 20%
* Patient with prior thoracic / abdominal radiotherapy for malignancy who was not discussed with sponsor before recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From randomisation up to 2 years of follow up
  Defined as the time from randomisation to the date of disease progression
Overall survival | From randomisation up to 2 years of follow up
  defined as the time from randomisation to the date of death from any cause.

SECONDARY OUTCOMES:
Number of PBT-related adverse events as assessed by CTCAE v5.0 | From start of PBT up to 2 years of follow up, for long term effects
  AEs related to proton beam therapy will be collected
The EORTC quality of life questionnaire (QLQ), EORTC QLQ-C30 score, scale of 0-100. | From randomisation up to 2 years of follow up
  Participant reported quality of life outcomes. The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / quality of life (QoL scale), and six single items. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
ED-5D-5L score | From randomisation up to 2 years of follow up
  Participant reported quality of life outcomes. The questionnaire comprises descriptive systems: mobility, self care, usual activities, pain/discomfort, anxiety/depression; scored from, level 1 to 5; level 1 indicating no problem and level 5 indicating unable to/extreme problems. There is also a scale from 0-100 to describe health status, 100 being the best health the patient can imagine, 0 being the worst health they can imagine.
Participant reported healthcare resource use from information collected on Client Service Receipt Inventory (CSRI) | From randomisation up to 2 years of follow up
  A tool used to collect participant reported information on the range of healthcare services and supports study participants may use, to calculate the rate of service usage to evaluate resource use as part of health economic analysis.
Measurement of costs in economic evaluations using iMTA Valuation of Informal Care (iVICQ) questionnaire | From randomisation up to 2 years of follow up
  Scoring (no scale) to evaluate health economics comparing PBT vs SOC surveillance and other SOC treatments for malignant pleural mesothelioma.

CONTACTS AND LOCATIONS:
Overall Officials: Crispin Hiley, Principal Investigator — University College, London
Locations (21):
- United Kingdom (21):
  - East Sussex Healthcare NHS Trust - Eastbourne Hospital, Eastbourne, East Sussex
  - East Sussex Healthcare NHS Trust - Conquest Hospital, Saint Leonards-on-Sea, East Sussex
  - Royal Berkshire Hospital, Reading, England
  - Southend University Hospital, Southend, Essex
  - Queen Alexandra Hospital, Portsmouth, Hampshire
  - Queen Elizabeth Hospital, King's Lynn, Kings Lynn, Norfolk
  - Betsi Cadwaladr University Health Board -Glan Clwyd Hospital, Bodelwyddan
  - Southmead Hospital, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Broomfield Hospital, Chelmsford
  - St James University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Clatterbridge Cancer Centre, Liverpool
  - St Bartholomew's Hospital, London
  - University College London Hospital, London
  - Maidstone Hospital, Maidstone
  - Christie Hospital, Manchester
  - Wythenshawe Hospital, Manchester
  - Weston Park Cancer Centre, Sheffield
  - Torbay Hospital, Torquay

IPD SHARING:
Plan to Share IPD: No